CLINICAL TRIAL: NCT07235839
Title: The Impact of an Advance Care Planning Game on Life-Sustaining Treatment Preferences, Depression, and Hope in Older Adults With Stroke
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lotung Poh-Ai Hospital (Other)
Responsible Party: Principal Investigator, Yu-Chun Chien, Principal Investigator, Lotung Poh-Ai Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IRB114-220-B
Record Dates: First submitted 2025-11-14; First posted 2025-11-19 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Stroke; Advance Care Planning
Keywords: stroke; Advance Care Planning; game; depression; hope
MeSH Terms: conditions — Stroke; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ACP Block Game Intervention (Experimental)
  Interventions: Other: ACP Block Game Intervention
- Usual Care (No Intervention): Routine stroke care

INTERVENTIONS:
Other: ACP Block Game Intervention — The "LOHAS Journey" Advance Care Planning (ACP) block game serves as an intervention. This non-invasive intervention, themed around a game-like journey, guides participants through various scenarios, allowing them to express their healthcare preferences through the blocks. The inclusion of "Hope Blocks" transforms several scenarios related to stroke and cancer, helping participants strengthen their hope for healthcare. The game also provides support tabs highlighting personal resources and potential future healthcare decision-makers. Beyond discussing life-sustaining treatment preferences, the game encourages expressing warm emotions such as gratitude and love.
  Arms: ACP Block Game Intervention

SUMMARY:
Stroke is the world's third leading cause of death and a major source of disability, with high rates of recurrence and mortality that often limit patients' ability to express their values and treatment preferences. This highlights the importance of Advance Care Planning (ACP) after stroke. This randomized controlled trial examined the effects of an ACP block-based game on life-sustaining treatment preferences, depression, and hope among adults aged 65-100 with subacute stroke in a regional teaching hospital. The Life Support Preferences Questionnaire (LSPQ) served as the primary outcome to assess preference changes immediately after the intervention and at four weeks, while the Hospital Anxiety and Depression Scale (HADS) and the Herth Hope Index (HHI) were secondary measures. The intervention used the "LOHAS Journey" ACP game, which applies travel-themed scenarios, blocks to express medical choices, hope-enhancing elements, and companion cards emphasizing personal resources and potential surrogate decision-makers, while also encouraging warm emotional expression. Generalized Estimating Equations (GEE) were used to analyze repeated measures and time-by-group effects. If effective, this ACP game may support broader clinical adoption of structured discussions on life-sustaining treatment preferences for older stroke patients.

DETAILED DESCRIPTION:
Background:

Stroke is the third leading cause of death worldwide and one of the most common causes of disability, accounting for approximately 10% of all deaths. One in four people experiences a stroke in their lifetime, and about 10% of stroke survivors face the risk of recurrent stroke within five years, often with more severe symptoms than the first episode. The one-year and five-year mortality rates after stroke are as high as 41% and 60%, respectively. Due to its high incidence, high recurrence rate, and high mortality, many stroke patients are unable to express their values and treatment preferences during the course of illness. This underscores the necessity of engaging in Advance Care Planning (ACP) discussions after stroke.

Purpose:

This study aims to explore the effects of an ACP game intervention on life-sustaining treatment preferences, depression, and hope among older adults with stroke.

Design:

A randomized controlled trial design was adopted.

Participants:

Using purposive sampling, we recruited subacute stroke patients aged 65-100 years from the neurology, neurosurgery, and rehabilitation wards of a regional teaching hospital in eastern Taiwan.

Measurement Tools:

The Life Support Preferences Questionnaire (LSPQ) was used as the primary outcome measure to assess differences in life-sustaining treatment preferences immediately after the intervention and at week 4 post-intervention. Secondary outcome measures included the Hospital Anxiety and Depression Scale (HADS) and the Herth Hope Index (HHI).

Intervention:

The intervention utilized the "LOHAS Journey" ACP block-based game developed for this study. The game incorporates travel-themed scenario guidance, allowing participants to express their medical preferences through the arrangement of blocks. "Hope blocks" were added to transform various stroke- and cancer-related scenarios, enhancing the participants' sense of hope. The game also includes companion option cards, emphasizing personal resources and potential future surrogate decision-makers. Beyond discussing life-sustaining treatment preferences, the game further encourages warm emotional expressions such as gratitude and affection.

Statistical Analysis:

Generalized Estimating Equations (GEE) were used to examine differences in life-sustaining treatment preferences, depression, and hope across repeated measurements, as well as to analyze time and group interaction effects.

If the effectiveness of the ACP block-based game on life-sustaining treatment preferences, depression, and hope among older adults with stroke is confirmed, it will support the promotion of ACP-related discussions in clinical stroke care.

ELIGIBILITY:
Inclusion Criteria:

* Older adults aged 65-100 years.
* Diagnosed with ischemic or hemorrhagic stroke confirmed by computer tomography (CT) or magnetic resonance imaging (MRI), and in the subacute stage 1-6 months after stroke onset.
* A National Institute of Health Stroke Scale (NIHSS) score ≤ 15, indicating mild to moderate stroke severity.
* Clear consciousness and able to communicate in Mandarin or Taiwanese.

Exclusion Criteria:

* Individuals diagnosed with chronic psychiatric disorders such as major depression, mania, or bipolar disorder.
* Older adults diagnosed with moderate to severe dementia.

Ages: 65 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2026-01-29 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
life support preferences questionnaire; LSPQ | From enrollment to the end of treatment at 5 weeks
  The questionnaire is designed to assess participants' preferences for various life-sustaining treatments across six medical scenarios and five treatment options. The maximum possible score is 150 and the minimum is 25. Higher scores indicate a greater willingness to receive life-sustaining medical treatments.

SECONDARY OUTCOMES:
hospital anxiety and depression scale; HADS | From enrollment to the end of treatment at 5 weeks
  This scale is used to screen for the prevalence of anxiety and depression among patients in medical settings who do not have psychiatric disorders. It contains 14 items, with a total score ranging from 0 to 21. Scores of 0-7 are considered within the normal range; scores of 8-10 indicate borderline or potential anxiety or depressive symptoms; and scores of ≥11 suggest the possible presence of emotional disorders or underlying conditions. Higher scores indicate more severe anxiety or depressive symptoms.
herth hope index; HHI | From enrollment to the end of treatment at 5 weeks
  This scale is used to assess the level of hope among patients with acute, chronic, or terminal illnesses. It consists of 12 items, with a total score ranging from 12 to 48. Higher scores indicate a higher level of hope.

CONTACTS AND LOCATIONS:
Locations (1):
- Lotong PohAi Hospital, Yilan, Taiwan

IPD SHARING:
Plan to Share IPD: No